CLINICAL TRIAL: NCT03637283
Title: Feasibility Study of Anti-VEGF Instead of Intraoperative Fan-shaped Photocoagulation in BRVO Combined With Vitreous Hemorrhage
Brief Title: Anti-VEGF Instead of Intraoperative Fan-shaped Photocoagulation in BRVO Combined With Vitreous Hemorrhage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Xiangtian Zhou, professor, Wenzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10008
Record Dates: First submitted 2018-08-15; First posted 2018-08-17 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Anti-VEGF; Branch Retinal Vein Occlusion; Vitrectomy
MeSH Terms: conditions — Retinal Vein Occlusion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anti-VEGF (Experimental): vitreoretinal surgery combined with intraoperative anti-VEGF
  Interventions: Procedure: anti-VEGF
- fan-shaped photocoagulation (Active Comparator): vitreoretinal surgery combined with fan-shaped photocoagulation
  Interventions: Procedure: fan-shaped photocoagulation

INTERVENTIONS:
Procedure: anti-VEGF — vitreoretinal surgery combined with intraoperative anti-VEGF
  Arms: anti-VEGF
Procedure: fan-shaped photocoagulation — vitreoretinal surgery combined with intraoperative fan-shaped photocoagulation
  Arms: fan-shaped photocoagulation

SUMMARY:
To evaluate the efficacy and safety of Anti-VEGF instead of intraoperative fan-shaped photocoagulation in BRVO combined with vitreous hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old;
2. BRVO is diagnosed
3. Vitreous hemorrhage
4. Vitreous hemorrhage combined with mild retinal fibrovascular proliferation (early fibrous vascular membrane, thin fibrous vascular membrane, loose retinal adhesion and intact local retinal structure)

Exclusion Criteria:

1. BRVO combined with severe retinal fibrovascular proliferation (long-term fibrovascular membrane, thick fibrous vascular membrane and tightly attached to the retina, deformation of local retinal, retinal tear or suspension of retinal vein )
2. BRVO combined with retinal detachment
3. Retinal veins are completely whitened
4. iris neovascularization or neovascular glaucoma
5. Combined glaucoma
6. combined with other retinopathy
7. Received anti-VEGF treatment within 3 months before surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in best-corrected visual acuity (BCVA) | 3 years
  Assessed using the ETDRS protocol

SECONDARY OUTCOMES:
Mean change from baseline in visual field | 3 years
  Assessed on Humphery(30-2 and 60-4)
chang from baseline in structure of retina | 3 years
  Assessed on Optical Coherence Tomography(OCT)
chang from baseline in retinal neovascularization | 3 years
  Assessed on Fundus Fluorescein Angiography(FFA)

CONTACTS AND LOCATIONS:
Overall Officials: Yong Wei, M.D, Principal Investigator — The Eye Hospital of Wenzhou Medical University